CLINICAL TRIAL: NCT03266094
Title: A Prospective, Multi-center, Single Arm Study of BiZact™ on Children and Adolescents Undergoing Tonsillectomy
Brief Title: A Study of BiZact™ on Children and Adolescents Undergoing Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT17024BZP
Record Dates: First submitted 2017-08-16; First posted 2017-08-29 (Actual); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Tonsillectomy
MeSH Terms: interventions — Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- A bipolar instrument for tonsillectomies (Other): A bipolar electrosurgical device that employs Radio frequency (RF) energy and pressure to ligate vessels interposed between its jaws which can then be transected using the built in knife deployed by the device trigger.
  Interventions: Device: BiZact™: A bipolar instrument for tonsillectomies

INTERVENTIONS:
Device: BiZact™: A bipolar instrument for tonsillectomies — A bipolar electrosurgical device that employs RF energy and pressure to ligate vessels interposed between its jaws which can then be transected using the built in knife deployed by the device trigger.

SUMMARY:
The purpose of this study is to assess safety and performance with the use of the BiZact™ device in tonsillectomy procedures in children and adolescents.

DETAILED DESCRIPTION:
A prospective, multi-center, single arm, study of BiZact™ on children and adolescents undergoing tonsillectomy.

Study Visits:

* Screening/Baseline
* Surgery, Day 0
* Post-Op Follow-up Day 1 - Day 7, Day 10, & Day 14 (Home assessments)
* Post-Op Follow-up Day 28 (Office Visit)

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescent subjects 2-12 years of age at the time of the procedure, inclusive
2. Scheduled to undergo tonsillectomy
3. The subject and subject's Legally Authorized Representative (LAR) is willing to participate and consents to participate, as documented by signed informed consent form and/ or assent form (as applicable)

Exclusion Criteria:

1. Subjects undergoing:

   1. Tonsillectomy as a result of cancer
   2. Unilateral tonsillectomy
2. Subjects with:

   1. Known Bleeding disorders
   2. History of peritonsillar abscess
   3. Craniofacial disorders
   4. Down's syndrome (Trisomy 21)
   5. Cerebral palsy
   6. Major heart disease (including but not limited to; right-sided heart failure, left-sided heart failure, congestive heart failure, coronary artery disease, arrhythmias, chronic heart failure, acute heart failure, etc.)
   7. Current tobacco use
3. Subjects unable to comply with the required study follow-up visits
4. Female subjects pregnant at time of procedure
5. The subject has comorbidities which, in the opinion of the Investigator, will not be appropriate for the study or the subject has an estimated life expectancy of less than 6 months.
6. The subject is participating or has participated in any drug or device research study within 30 days of enrollment.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Brown, MD, Principal Investigator — Coastal Pediatric Research
Locations (2):
- United States (2):
  - Southeast Clinical Research Associates, LLC, Charlotte, North Carolina
  - Coastal Pediatric Associates, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 children, ages 2 to 12 in the US, were enrolled into a single-arm trial. A total of 60 subjects were screened and consented.
Groups:
- BiZact Arm: A bipolar electrosurgical device that employs Radio frequency (RF) energy and pressure to ligate vessels interposed between its jaws which can then be transected using the built in knife deployed by the device trigger.
Period: Overall Study
Arm/Group | BiZact Arm
Started | 60
Completed | 58
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: During the study, 60 patients were screened, and 60 patients were consented and enrolled in the study. One patient was lost to follow-up. Another patient withdrew from the study during post-procedure follow-up. Both patients were still included in the intent-to-treat data analysis with the data obtained.
Groups:
- BiZact Arm: 60 Pediatric subjects undergoing tonsillectomy
Arm/Group | BiZact Arm
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.7 (2.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60
Undergoing Tonsillectomy [Count of Participants; unit: Participants] | 60
Signed Informed Consent [Count of Participants; unit: Participants] | 60

OUTCOME MEASURES:

1. Primary Outcome: Intra-operative Blood Loss
Description: The study will be considered a success if the mean intra-operative blood loss is less than the mean intra-operative blood loss associated with conventional tonsillectomy in a large meta-analysis
Time Frame: During procedure
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | A Bipolar Instrument for Tonsillectomies
Number analyzed (Participants) | 60
mL | 1.7 (2.38)

2. Primary Outcome: Number of Patients With Intra-operative Blood Loss
Description: as for outcome 1
Time Frame: During procedure
Population: Intra-operative bleeding occurred in 29 of the 60 patients. For subjects with no intra-operative bleeding, volume was considered as 0 mL.
Measure: Count of Participants; unit: Participants
Groups:
- A Bipolar Instrument for Tonsillectomies: A bipolar electrosurgical device that employs RF energy and pressure to ligate vessels interposed between its jaws which can then be transected using the built in knife deployed by the device trigger.
  BiZact™: A bipolar instrument for tonsillectomies: A bipolar electrosurgical device that employs RF energy and pressure to ligate vessels interposed between its jaws which can then be transected using the built in knife deployed by the device trigger.
Arm/Group | A Bipolar Instrument for Tonsillectomies
Number analyzed (Participants) | 29
Participants
  Patients with Intra-operative bleeding | 29
  Patients age 3-5 | 9
  Patients age 6-12 | 20

3. Secondary Outcome: Number of Cases/Participants Rated Under Different Categories Based on the Performance of the Investigational Device
Description: Ability to dissect tonsils with investigational device via Likert Scale (Very Good, Good, Acceptable, Poor, Very Poor).
Time Frame: During Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | A Bipolar Instrument for Tonsillectomies
Number analyzed (Participants) | 60
Participants
  Very Good | 51
  Good | 6
  Acceptable | 1
  Poor | 1
  Very Poor | 1

4. Secondary Outcome: Number of Cases With Ability to Achieve Hemostasis (Performance of the Investigational Device)
Description: Ability to achieve hemostasis (arrest of bleeding, as assessed by visual inspection of the Investigator) without the use of other interventions (e.g. energy device or sutures)
Time Frame: During Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | A Bipolar Instrument for Tonsillectomies
Number analyzed (Participants) | 60
Participants | 60

5. Secondary Outcome: "Number of Cases/Participants With Analgesic Consumption
Description: Analgesic consumption (standard of care) and concomitant medications (via patient diary).
Time Frame: 28 days post-operatively
Population: Caregivers were instructed to complete the take-home diary and record analgesics given on days 1-6, 7, 10, 14, and 28. Compliance with completing the diaries was not 100% and therefore we do not have data for all 60 subjects. Missing data was recorded as a protocol deviation.
Measure: Count of Participants; unit: Participants
Arm/Group | A Bipolar Instrument for Tonsillectomies
Number analyzed (Participants) | 60
Participants
  Day 0 | 58
  Day 1: number analyzed (Participants) | 58
  Day 1 | 56
  Day 2: number analyzed (Participants) | 58
  Day 2 | 55
  Day 3: number analyzed (Participants) | 58
  Day 3 | 54
  Day 4: number analyzed (Participants) | 58
  Day 4 | 53
  Day 5: number analyzed (Participants) | 58
  Day 5 | 49
  Day 6: number analyzed (Participants) | 57
  Day 6 | 49
  Day 7: number analyzed (Participants) | 53
  Day 7 | 44
  Day 10: number analyzed (Participants) | 57
  Day 10 | 19
  Day 14: number analyzed (Participants) | 56
  Day 14 | 6
  Day 28: number analyzed (Participants) | 57
  Day 28 | 1

6. Secondary Outcome: Post-operative Pain
Description: Evaluation of post-operative pain incidence and severity measured using the Wong-Baker FACES® Pain Rating Scale, an illustrated pain scale ranging from a happy face at 0 "No Hurt" to a crying face at 10 "Hurts Worst".
Time Frame: Post-operative Day 4
Population: Post-operative pain levels were collected via patient diaries provided for the caregiver to complete. Only 58 caregivers completed the diary for day 4, so only 58 participants were included in the analysis. The missed days of data collection were recorded as protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 58
score on a scale | 4.7 (2.93)

7. Secondary Outcome: Post-operative Pain
Description: as for outcome 6
Time Frame: Post-operative Day 5
Population: Post-operative pain levels were collected via patient diaries provided for the caregiver to complete. Only 58 caregivers completed the diary for day 5, so only 58 participants were included in the analysis. The missed days of data collection were recorded as protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 58
score on a scale | 4.5 (2.79)

8. Secondary Outcome: Post-operative Pain
Description: as for outcome 6
Time Frame: Post-operative Day 6
Population: Post-operative pain levels were collected via patient diaries provided for the caregiver to complete. Only 57 caregivers completed the diary for day 6, so only 57 participants were included in the analysis. The missed days of data collection were recorded as protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 57
score on a scale | 3.7 (2.61)

9. Secondary Outcome: Post-operative Pain
Description: as for outcome 6
Time Frame: Post-operative Day 7
Population: Post-operative pain levels were collected via patient diaries provided for the caregiver to complete. Only 53 caregivers completed the diary for day 7, so only 53 participants were included in the analysis. The missed days of data collection were recorded as protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 53
score on a scale | 3.3 (2.83)

10. Secondary Outcome: Post-operative Pain
Description: as for outcome 6
Time Frame: Post-operative Day 10
Population: Post-operative pain levels were collected via patient diaries provided for the caregiver to complete. Only 57 caregivers completed the diary for day 10, so only 57 participants were included in the analysis. The missed days of data collection were recorded as protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 57
score on a scale | 1.5 (2.16)

11. Secondary Outcome: Post-operative Pain
Description: as for outcome 6
Time Frame: Post-operative Day 14
Population: Post-operative pain levels were collected via patient diaries provided for the caregiver to complete. Only 56 caregivers completed the diary for day 14, so only 56 participants were included in the analysis. The missed days of data collection were recorded as protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 56
score on a scale | 0.8 (1.82)

12. Secondary Outcome: Post-operative Pain
Description: as for outcome 6
Time Frame: Post-operative Day 28
Population: Post-operative pain levels were collected via patient diaries provided for the caregiver to complete. Only 57 caregivers completed the diary for day 28, so only 57 participants were included in the analysis. The missed days of data collection were recorded as protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 57
score on a scale | 0.3 (1.18)

13. Secondary Outcome: Post-operative Pain
Description: as for outcome 6
Time Frame: Day 1
Population: Post-operative pain levels were collected via patient diaries provided for the caregiver to complete. Only 58 caregivers completed the diary for day 1, so only 58 participants were included in the analysis. The missed days of data collection were recorded as protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 58
score on a scale | 5.4 (2.94)

14. Secondary Outcome: Post-operative Pain
Description: as for outcome 6
Time Frame: Day 2
Population: Post-operative pain levels were collected via patient diaries provided for the caregiver to complete. Only 58 caregivers completed the diary for day 2, so only 58 participants were included in the analysis. The missed days of data collection were recorded as protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 58
score on a scale | 5.1 (2.83)

15. Secondary Outcome: Post-operative Pain
Description: as for outcome 6
Time Frame: Day 3
Population: Post-operative pain levels were collected via patient diaries provided for the caregiver to complete. Only 58 caregivers completed the diary for day 3, so only 58 participants were included in the analysis. The missed days of data collection were recorded as protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiZact Arm
Number analyzed (Participants) | 58
score on a scale | 4.9 (2.83)

ADVERSE EVENTS:
Time Frame: Day 0 (after commencement of surgery with BiZact™ to 28 (+7) days follow-up
Description: Definition of adverse event is consistent with clinicaltrials.gov.
  The relationship to the study-device was "not related" for 100% of Adverse Event (AE) reports. There have been no serious adverse events, unanticipated adverse device effects, unanticipated serious adverse device effects reported in the study.
Arm/Group | BiZact Arm
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 27/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BiZact Arm (N=60)
Right Knee Injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Fever (Infections and infestations) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Influenza (Infections and infestations) | 3 (3)
Swollen Tongue (Injury, poisoning and procedural complications) | 2 (2)
Cold (Infections and infestations) | 1 (1)
Headache (Infections and infestations) | 2 (2)
Viral Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Head Laceration (Injury, poisoning and procedural complications) | 1 (1)
Bilateral Inferior Turbinate Hypertrophy (Ear and labyrinth disorders) | 1 (1)
Cough (Infections and infestations) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 4 (4)
Strep Throat (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Dehydration (Injury, poisoning and procedural complications) | 4 (5)
Significant Pain in Throat (Injury, poisoning and procedural complications) | 2 (2)
Ear Infection (Infections and infestations) | 1 (1)
Epistaxis (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT03266094/Prot_SAP_000.pdf